CLINICAL TRIAL: NCT00503646
Title: Communication and Intimacy-Enhancing Intervention for Men Diagnosed With Early Stage Prostate Cancer and Their Partners: A Pilot and Feasibility Trial
Brief Title: Communication and Intimacy-Enhancing Therapy for Men With Early Stage Prostate Cancer and Their Partners
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized
Other Study IDs: 07-069; MSKCC-07069
Record Dates: First submitted 2007-07-17; First posted 2007-07-19 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2009-07

CONDITIONS: Prostate Cancer; Psychosocial Effects of Cancer and Its Treatment; Sexual Dysfunction and Infertility; Sexuality and Reproductive Issues
Keywords: psychosocial effects of cancer and its treatment; sexual dysfunction and infertility; sexuality and reproductive issues; stage IIB prostate cancer; stage IIA prostate cancer; stage I prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms; Sexual Dysfunction, Physiological; Infertility; Sexuality | interventions — Counseling; Psychiatric Rehabilitation

INTERVENTIONS:
Other: communication intervention
Other: counseling intervention
Other: questionnaire administration
Procedure: psychosocial assessment and care

SUMMARY:
RATIONALE: Participating in a therapy program may enhance communication and intimacy between men with prostate cancer and their partners.

PURPOSE: This randomized clinical trial is studying how well therapy enhances communication and intimacy for men with early stage prostate cancer and for their partners.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the feasibility and acceptability of conducting a randomized clinical trial evaluating communication and intimacy-enhancing intervention (CI) vs usual care (UC).
* To collect descriptive information and basic psychometrics on proposed study measures.
* To gather preliminary data regarding the impact of CI on couples' psychosocial adaptation, relationship closeness, and sexual intimacy in order to calculate power for a larger full scale trial.

OUTLINE: This is a multicenter study. Patients and their partners are randomized to 1 of 2 intervention arms.

* Arm I: Patients and their partners receive communication and intimacy-enhancing intervention (CI) once a week comprising the following five 90-minute sessions: Rationale and Overview; Basic Communication; Intimacy and Sexuality; Improving Intimacy; and Reflecting on Changes and Cancer Survivorship.
* Arm II: Patients and their partners receive standard psychological and emotional care (usual care [UC]) (i.e., social work consultations and referral to a psychiatrist or psychologist, if requested or deemed necessary by the attending physician).

Physical impairment, psychological adjustment, relationship closeness, relationship communication, sexual function and satisfaction, male self-esteem, relationship satisfaction, intervention evaluation, and erectile dysfunction treatment utilization, and referral are assessed at 1 week post-intervention or at 6-8 weeks post baseline and then at 3 months (for patients and their partners in arm I) and at 8 weeks post-baseline and then at 3 months (for patients and their partners in arm II).

PROJECTED ACCRUAL: A total of 50 patients and 50 partners will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Patient has a primary diagnosis of localized (early stage) prostate cancer

  * Has undergone surgery within the past year
* Patient and partner married or cohabiting and relationship duration ≥ 1 year

PATIENT CHARACTERISTICS:

* ECOG performance status 0 or 1 at the time of initial recruitment
* Lives within 2-hour commuting distance from recruitment center (MSKCC or FCCC)
* No significant self-identified hearing impairment that would preclude study participation

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-05; Primary Completion 2010-05 (Estimated)

PRIMARY OUTCOMES:
Feasibility and acceptability
Descriptive characteristics of study measures
Impact of communication intervention on couples' psychological adaptation, relationship closeness, and sexual intimacy

CONTACTS AND LOCATIONS:
Overall Officials: David W. Kissane, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Christian J. Nelson, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania

REFERENCES:
- [Result] Manne S, Badr H, Zaider T, Nelson C, Kissane D. Cancer-related communication, relationship intimacy, and psychological distress among couples coping with localized prostate cancer. J Cancer Surviv. 2010 Mar;4(1):74-85. doi: 10.1007/s11764-009-0109-y. Epub 2009 Dec 6. PMID 19967408